CLINICAL TRIAL: NCT01407666
Title: Prospective Randomized Comparative Study Between Epidural and Bilateral Paravertebral Blocks for Perioperative Pain Management in Patients Undergoing Open Liver Resection
Brief Title: Comparison Between Epidural and Bilateral Paravertebral Blocks in Liver Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOD09070393-01 / PRO09070393
Record Dates: First submitted 2011-02-17; First posted 2011-08-02 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Liver Disease; Pain
Keywords: paravertebral block; epidural block; pain management; liver resection; comparison
MeSH Terms: conditions — Liver Diseases; Pain; Agnosia | interventions — Anesthesia, Conduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bilateral paravertebral blocks (Experimental): Bilateral continuous paravertebral blocks for open liver resection
  Interventions: Procedure: paravertebral blocks
- epidural block (No Intervention): received thoracic epidural block for open liver resection

INTERVENTIONS:
Procedure: paravertebral blocks — use bilateral thoracic paravertebral blocks for pain control
  Other Names: regional anesthesia
  Arms: Bilateral paravertebral blocks

SUMMARY:
This prospective, randomized study is intended to assess the efficacy and safety of bilateral continuous paravertebral blocks compared to continuous epidural block for open liver resection. Hypotheses: Bilateral paravertebral blocks are: 1) equally effective in controlling the perioperative pain; and 2) safe, with less frequent complications following open liver resection when compared to continuous epidural block.

DETAILED DESCRIPTION:
Background: A number of studies evaluating unilateral continuous paravertebral block demonstrate equal or superior analgesia when compared to epidural analgesia for postoperative pain control (1-7). At the same time, these studies show a decreased incidence of side effects and complications, including: hypotension, pulmonary complications, urinary retention, nausea and vomiting and failed blocks. Several studies also indicate that bilateral paravertebral blocks provide adequate postoperative analgesia (8-14). However, no study has been performed to date that shows a direct comparison between epidural and bilateral paravertebral blocks in patients undergoing open liver resection.Objectives: This prospective, randomized study is intended to assess the efficacy and safety of bilateral continuous paravertebral blocks compared to continuous epidural block for open liver resection. Hypotheses: Bilateral paravertebral blocks are: 1) equally effective in controlling the perioperative pain; and 2) safe, with less frequent complications following open liver resection when compared to continuous epidural block.Methods: A hundred adult patients undergoing elective open liver resection will be randomized to receive a continuous epidural block or continuous bilateral paravertebral blocks for perioperative analgesia. The primary outcome will be the degree of pain control measured by visual analog scale at 24 hours post surgery (at rest and while the patient is performing maximum incentive spirometry). The secondary outcomes will include: 1) Assessment of pain (at rest, with cough, and with ambulation) using the verbal numerical pain scale will be performed postoperatively every 8 hours by floor nursing staff until discharge. During the night the patient will not be awakened for pain assessment. 2) Intravenous opioid requirement: In addition to pain score, postoperative intravenous opioid requirements [hydromorphone (mg)] will also be recorded daily; Frequency of side effects and complications; and other functional status (volume of maximum incentive spirometry, time to extubation, total time for initial ambulation, the length of the hospital stay, time to return of bowel function, readiness for discharge from the hospital, and length of hospital stay). At one month post surgery, health-related quality of life, mortality, and any morbidities will be assessed. Each variable will be compared between the paravertebral group and the epidural group to examine the hypotheses above. Clinical Implications: Bilateral continuous paravertebral blocks could be an equally effective and safe alternative to a continuous epidural block for perioperative pain management in patients who undergo open liver resection.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status (ASAPS) I to III patients aged over 18 years and scheduled to undergo elective open liver resection at UPMC Presbyterian/Montefiore Hospital will be screened for enrollment in the study. One hundred (100) patients will be enrolled in this study with equal numbers (n = 50) in each arm of the trial. In order to avoid skewed sex difference between the two groups, the sex will be allocated.

Exclusion Criteria:

* non elective surgery,
* ASAPS IV or greater,
* age younger than 18 years,
* any contraindication to the placement of an epidural catheter or bilateral paravertebral catheters
* chronic pain conditions
* preoperative opioid use
* coagulation abnormalities or patients who are expected to be on therapeutic anticoagulants postoperatively
* allergy to any of the drugs/agents used our study protocol
* preoperative chronic renal dysfunction, who requires renal replacement therapy or serum creatinine greater than 1.4 mg/dL
* altered mental status (not oriented to place, person, or time),
* any comorbid conditions that, in the judgment of the consulting surgeon or anesthesiologist, would proscribe the patient from any aspect of the study, -
* inability to provide adequate informed consent
* refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-08; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Pain immediately after maximum incentive spirometry | 24 hours postoperatively
  Pain will be assessed using an 11-point verbal numerical pain scale (VAS) with 0 indicating no pain and 10 indicating the worst pain imaginable;(21) pain will be determined 24 hours postoperatively immediately after maximum incentive spirometry.

SECONDARY OUTCOMES:
date of the removal of the catheter | up to one week after the surgery
  date of the removal of the catheter with any requirement of blood transfusion because of coagulation

CONTACTS AND LOCATIONS:
Overall Officials: Tetsuro Sakai, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania, United States